CLINICAL TRIAL: NCT06041802
Title: A Phase 2 Clinical Study to Evaluate the Safety and Efficacy of MK-3475A in Japanese Participants With Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (R/M cSCC) or Locally Advanced (LA) Unresectable cSCC.
Brief Title: A Study of Pembrolizumab (+) Berahyaluronidase Alfa (MK-3475A) (Pembrolizumab Formulated With Berahyaluronidase Alfa (MK-5180)) in Japanese Participants With Recurrent or Metastatic Cutaneous Squamous Cell Carcinoma (R/M cSCC) or Locally Advanced (LA) Unresectable cSCC (MK-3475A-E39)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-E39; MK-3475A-E39 (Other: MSD); jRCT2041230074 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Squamous Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (+) Berahyaluronidase alfa (Experimental): Participants will receive pembrolizumab (+) berahyaluronidase alfa subcutaneously for up to 18 administrations.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Pembrolizumab (+) Berahyaluronidase alfa is a fixed-dose formulation of pembrolizumab and berahyaluronidase alfa for SC administration.
  Other Names: MK-3475A

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of subcutaneous (SC) pembrolizumab (+) berahyaluronidase alfa in Japanese participants with recurrent or metastatic cutaneous squamous cell carcinoma or locally advanced unresectable cSCC. The primary hypothesis is that pembrolizumab (+) berahyaluronidase alfa will result in greater than 10% objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR).

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically confirmed cSCC by the investigator as the primary site of malignancy
* R/M cSCC cohort only: Has metastatic disease, defined as disseminated disease distant to the initial/primary site of diagnosis, and/or has locally recurrent disease that has been previously treated (with either surgery or radiotherapy) and is not curable by either surgery or radiotherapy
* LA unresectable cSCC cohort only: Is ineligible for surgical resection
* LA unresectable cSCC cohort only: Has received prior radiation therapy (RT) to index site or has been deemed to be not eligible for RT
* LA unresectable cSCC cohort only: Has received prior systemic therapy for curative intent are eligible regardless of regimen
* Has a life expectancy of greater than 3 months
* Must provide archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated

Exclusion Criteria:

* Has cSCC that can be cured with surgical resection, radiotherapy, or with a combination of surgery and radiotherapy.
* Has any other histologic type of skin cancer other than invasive squamous cell carcinoma as the primary disease under study
* Has received prior systemic anticancer therapy including investigation agents within 4 weeks before allocation
* Has not adequately recovered from major surgery or has ongoing surgical complications
* Received prior radiotherapy within 2 weeks of study intervention, or had radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has an ongoing active infection requiring systemic therapy
* Has a history of human immunodeficiency virus (HIV) infection
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has history of allogenic tissue/organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 40 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 40 months
  For participants who demonstrate CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Disease Control Rate (DCR) | Up to approximately 40 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who demonstrate a confirmed CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.]).The DCR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 40 months
  OS is defined as the time from first dose of study treatment to death due to any cause.
Number of Participants who Experience an Adverse Event (AE) | Up to approximately 28 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience at least one AE will be reported.
Number of Participants who Discontinue Due to an AE | Up to approximately 25 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (18):
- Japan (18):
  - Nagoya University Hospital ( Site 0003), Nagoya, Aichi-ken
  - Sapporo Medical University Hospital ( Site 0002), Sapporo, Hokkaido
  - Yokohama City University Hospital ( Site 0016), Yokohama, Kanagawa
  - Tohoku University Hospital ( Site 0019), Sendai, Miyagi
  - Shinshu University Hospital ( Site 0011), Matsumoto, Nagano
  - Niigata Cancer Center Hospital ( Site 0005), Niigata, Niigata
  - Saitama Medical University International Medical Center ( Site 0008), Hidaka, Saitama
  - Shimane University Hospital ( Site 0014), Izumo, Shimane
  - Shizuoka Cancer Center ( Site 0004), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 0007), Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 0018), Koto, Tokyo
  - Chiba University Hospital ( Site 0001), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0017), Fukuoka
  - National Hospital Organization Kagoshima Medical Center ( Site 0013), Kagoshima
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 0012), Kyoto
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 0009), Osaka
  - Keio University Hospital ( Site 0010), Tokyo
  - Wakayama Medical University Hospital ( Site 0015), Wakayama

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/